CLINICAL TRIAL: NCT05517239
Title: Phase II Study of Gemcitabine With Oxaliplatin in Patients With Advanced Hepatocellular Carcinoma After Failure of Sorafenib Treatment
Brief Title: Gemcitabine With Oxaliplatin (GEMOX) in Patients With Advanced Hepatocellular Carcinoma After Failure of Sorafenib Treatment
Acronym: PEACH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0269
Record Dates: First submitted 2022-08-08; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma, Unresectable, Advanced
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — gemcitabine-oxaliplatin regimen; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine, Oxaliplatin (Experimental): Gemcitabine 1,000 mg/m2 infusion for 30minutes and followed by oxaliplatin 100mg/m2 infusion for 2hours on day1. All drugs were administered intravenously until progression, intolerance, patient withdrawal, or death.
  Interventions: Drug: Gemcitabine, Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine, Oxaliplatin — Gemcitabine 1,000 mg/m2 infusion for 30minutes and followed by oxaliplatin 100mg/m2 infusion for 2hours on day1. All drugs were administered intravenously until progression, intolerance, patient withdrawal, or death.
  Other Names: Gemzar, Eloxatin

SUMMARY:
The purpose of this study is to test the safety of gemcitabine and oxaliplatin regimen and to see its effects on sorafenib treatment failed hepatocellular carcinoma patients.

DETAILED DESCRIPTION:
Patients who progressed after or cannot tolerate sorafenib treatment. Patients who cannot receive sorafenib for other reason are also permitted. Treatment is given in cycles, each cycle is 2 weeks long. Tumor measurements by CT and/or MRI will be repeated every 3 cycles. Patients will continue to receive study treatment as long as there is no disease progression or unacceptable side affects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who signed informed consent.
2. Male or female ≥ 20 years of age.
3. Diagnosis of advanced HCC according to the AASLD.
4. Unresectable HCC
5. Advanced disease defined as extrahepatic metastasis or locally advanced disease not amenable to surgical resection or other local-regional therapies including transhepatic arterial (chemo) embolization (TACE or TAE) and local ablative therapy
6. Patient who progressed after prior local-regional therapy (local-regional therapy must be completed at least 4weeks prior to the baseline).
7. Patients who progressed after or cannot tolerate sorafenib treatment. Patients who cannot receive sorafenib for other reason are also permitted.

   * Documented radiological confirmation of disease progression during or after sorafenib treatment
   * Intolerance to sorafenib is defined as documented sorafenib-related grade 3 or 4 adverse events that led to sorafenib discontinuation
8. Patients must have a life expectancy of at least 12 weeks.
9. Eastern Cooperative Oncology Group (ECOG) performance state ≤ 2
10. Measurable lesion according to the RECIST 1.1 criteria
11. Child Pugh Class A or B7
12. Patients must have adequate organ and marrow function:

    * Absolute neutrophil count (ANC) ≥1.5X10^9/L
    * Platelets≥75X10^9/L
    * Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) < 5 Upper Normal Limit(UNL)
    * Total Bilirubin≤1.5 X UNL
13. Controlled brain metastasis is allowed(except brain metastasis to require treatment to control symptom-wash out of treatment for brain metastasis is not required.)

Exclusion Criteria:

1. Imaging findings for HCC corresponding to any of the following

   * HCC with >60% liver occupation
   * Portal vein invasion at the main portal branch (Vp4)
2. History of a secondary malignancy within 3 years

   - in situ cervical cancer, adequately treated basal cell or superficial bladder cancer
3. History of chemotherapy or radiotherapy within 4 weeks

   - but, 2 weeks for sorafenib and radiotherapy site of bone lesion
4. Patient who not recovered toxicity ≥ grade 2 related prior local-regional therapy or systemic therapy.
5. Patients with any known severe allergy to Gemcitabine or platinum compound.
6. Active gastro-Intestinal bleeding.
7. Patients who are receiving any other chemotherapy or study treatments.
8. Pregnant or lactating women or women of childbearing potential without proper contraceptive methods.
9. Patients with active infections requiring an IV antibiotic.
10. Neuropathy ≥ grade 2
11. Patients with known interstitial lung disease or pulmonary fibrosis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 1 year
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From enrollment to 30 days follow-up after the end of treatment
  Overall safety profile verified as relevance of adverse events and laboratory abnormality based on CTCAE v4.0.
Response rate | from enrollment to 1 year follow-up after the end of treatment
  Assessed by RECIST 1.1
Overall survival | From enrollment to 1 year follow-up after the end of treatment
  Estimated by the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Hye Jin Choi, Principal Investigator — Division of Medical Oncology, Department of Internal Medicine, Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No